CLINICAL TRIAL: NCT02127658
Title: MRSA Eradication and Decolonization in Children
Acronym: MEDiC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit all planned participants prior to end of funding
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Paul Musey, Assistant Professor of Clinical Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R24HS022434-01, 1305011439; 1R24HS022434-01 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-05

CONDITIONS: MRSA
MeSH Terms: interventions — Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hygiene education (Active Comparator): Participants will receive specific hygiene instructions according to existing recommendations from the Ryan White Center for Pediatric Infectious Disease, Riley Hospital.
  Interventions: Other: Hygiene education
- Hygiene education and Decolonization (Active Comparator): Participants in this intervention group will receive the same hygiene instructions as the participants in the first intervention group. In addition, intervention number 2 will include the following for all consented household members: Twice weekly 15 minute soaks in diluted bleach water (2/3 cup of 8.25% sodium hypochlorite [Clorox; The Clorox Company] for a standard 50 gallon tub of water, or a teaspoon for each 1.5 gallons of water used) for the duration of 6 weeks. Application of 2% mupirocin ointment by the use of clean swab to the bilateral anterior nares twice daily for ten days
  Interventions: Other: Sodium Hypochlorite; Drug: Mupirocin ointment

INTERVENTIONS:
Other: Hygiene education — Participants will receive specific hygiene instructions according to existing recommendations.
  Arms: Hygiene education
Other: Sodium Hypochlorite — Participants in this intervention group will receive the same hygiene instructions as the participants in the first intervention group. In addition, intervention number 2 will include the following for all consented household members: Twice weekly 15 minute soaks in diluted bleach water (2/3 cup of 8.25% sodium hypochlorite [Clorox; The Clorox Company] for a standard 50 gallon tub of water, or a teaspoon for each 1.5 gallons of water used) for the duration of 6 weeks. Application of 2% mupirocin ointment by the use of clean swab to the bilateral anterior nares twice daily for ten days
  Arms: Hygiene education and Decolonization
Drug: Mupirocin ointment — Participants in this intervention group will receive the same hygiene instructions as the participants in the first intervention group. In addition, intervention number 2 will include the following for all consented household members: Twice weekly 15 minute soaks in diluted bleach water (2/3 cup of 8.25% sodium hypochlorite [Clorox; The Clorox Company] for a standard 50 gallon tub of water, or a teaspoon for each 1.5 gallons of water used) for the duration of 6 weeks. Application of 2% mupirocin ointment by the use of clean swab to the bilateral anterior nares twice daily for ten days
  Arms: Hygiene education and Decolonization

SUMMARY:
In this study, the investigators intend to compare therapies (abscess surgery and hygiene education compared to abscess surgery and hygiene education followed by decolonization) for Methicillin-Resistant Staphylococcus Aureus skin and soft tissue infections (MRSA SSTI) to determine which is the more effective treatment. The investigators focus on patient centered outcomes as described by the families of MRSA infected patients. Such outcomes are likely to include quality of life, side effects, and school and work attendance. The hypothesis is that treatment with decolonization will decrease the rate of SSTI recurrence and improve overall patient centered outcomes. The rationale is that negative outcomes such as recurrence may be avoided through the use of readily available prevention strategies, but that it is important to determine how burdensome those prevention strategies are for patients and families.

DETAILED DESCRIPTION:
The past two decades have seen a dramatic increase in skin and soft tissue infections (SSTI) caused by antibiotic resistant bacteria Methicillin-resistant Staphylococcus aureus (MRSA). The shift from hospital-acquired infections to community-acquired infections has resulted in many otherwise healthy children being affected. Recent estimates are that the US incidence of hospitalizations caused by MRSA SSTI is > 45 per 100,000 children, with many children requiring surgical procedures to drain pus caused by the infection.

Treatment of MRSA SSTI usually involves abscess surgery (incision and drainage), but recurrence of infection can be as high as 72%. Decolonization protocols are, therefore, sometimes recommended to eradicate the bacteria and decrease recurrence. These measures can be burdensome for the patient, consisting of regular bleach baths or chlorhexidine body washes, and/or daily nasal antibiotics. The Infectious Disease Society of America supports decolonization, but acknowledges that the recommendations are based on limited, non-MRSA specific data. One small, randomized controlled trial of children with Staphylococcus aureus infection (MRSA and non MRSA) has shown a short lasting effect (4 months) on skin colonization (presence of bacteria on the skin), and an even shorter lasting effect (1 month) on SSTI recurrence. The effect of decolonization on patient-centered outcomes such as quality of life and school attendance has not been assessed.

In this study, the investigators intend to compare therapies (abscess surgery and hygiene education compared to abscess surgery and hygiene education followed by decolonization) for Methicillin-Resistant Staphylococcus Aureus skin and soft tissue infections (MRSA SSTI) to determine which is the more effective treatment. The investigators focus on patient centered outcomes as described by the families of MRSA infected patients. Such outcomes are likely to include quality of life, side effects, and school and work attendance. The hypothesis is that treatment with decolonization will decrease the rate of SSTI recurrence and improve overall patient centered outcomes. The rationale is that negative outcomes such as recurrence may be avoided through the use of readily available prevention strategies, but that it is important to determine how burdensome those prevention strategies are for patients and families.

ELIGIBILITY:
Inclusion Criteria:

* Children/youth ages 3 months - 18 years seen in the Riley Pediatric Surgery Outpatient Clinic for a follow up visit within two weeks of the incision and drainage of a culture-confirmed MRSA abscess (regardless of where the abscess was drained)
* Children/youth ages 3 months - 18 years who had an incision and drainage of a culture-confirmed MRSA abscess in the Riley Emergency Department or Riley Operating Room within the two weeks prior to enrollment
* Household members of the patient who are between the ages 3 months - 64 years

Exclusion Criteria:

* Children in need of additional abscess surgery
* Documented immune deficiency
* Previous burn victims
* Self reported history of sensitivity to chlorine bleach or mupirocin
* Families without a bathtub

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul I Musey, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Pediatric Surgery Outpatient Clinic, Riley Outpatient Center, Riley Hospital for Children, Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore CM, Wiehe SE, Lynch DO, Claxton GE, Landman MP, Carroll AE, Musey PI. Methicillin-Resistant Staphylococcus aureus Eradication and Decolonization in Children Study (Part 1): Development of a Decolonization Toolkit With Patient and Parent Advisors. J Particip Med. 2020 May 20;12(2):e14974. doi: 10.2196/14974. PMID 33064109
- [Derived] Moore CM, Wiehe SE, Lynch DO, Claxton GE, Landman MP, Carroll AE, Musey PI. Methicillin-Resistant Staphylococcus aureus Eradication and Decolonization in Children Study (Part 2): Patient- and Parent-Centered Outcomes of Decolonization. J Particip Med. 2020 May 20;12(2):e14973. doi: 10.2196/14973. PMID 33064098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In-person recruitment will be done in the pediatric surgery outpatient clinic located in the Riley Outpatient Center Riley Hospital for Children, Indiana University Health, Indianapolis, Indiana. Recruitment will also be done via phone for patients who had an incision and draining procedure of a culture-confirmed Methicillin-Resistant Staphylococcus Aureus (MRSA) abscess in the Riley Emergency Department (ED), Riley Operating Room (OR), or IU Health North Operating Room (OR).
Groups:
- Hygiene Education: Participants will receive specific hygiene instructions according to existing recommendations from the Ryan White Center for Pediatric Infectious Disease, Riley Hospital as outlined here:
  * Take daily showers or bath with soap
  * Clean hands with soap and water or with hand sanitizers when hands are dirty, and after each bathroom break or diaper change
  * Don't share towels, wash cloths, clothing, toothbrushes, or razors within the family or with friends
  * Discard lotions in jars (can be easily contaminated with MRSA when someone puts their hand in a jar)
  * Keep all wounds including cuts and scrapes clean and covered until healed
  * Avoid other person's dirty bandages or uncovered wounds
  * Encourage athletes or health club members to shower before and after all practices and competitions, and wipe down equipment surfaces before and after use
  * Uniforms and practice jerseys should be washed after each game or practice. Sports equipment should be washed/cleaned weekly
  * Wash all towels, wash cloths, sleepwear, underwear, and linens in hot water with laundry detergent once weekly and dry with hot air in a dryer
Period: Overall Study
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Started | 7 | 7
6 Week Follow-up | 5 | 4
6 Month Follow-up | 5 | 3
12 Month Follow-up | 5 | 2
Completed | 5 | 4
Not Completed | 2 | 3
Not completed — Screen Fail (Not MRSA on culture check) | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hygiene Education | Hygiene Education and Decolonization | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.6 (2.81) | 3.5 (4.67) | 3.5 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 3 | 6
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 0 | 2
Surgical Drainage procedure location [Count of Participants; unit: Participants] — Where the incision and drainage procedure took place (Operating room vs Emergency Department).
  Participants
    Operating Room | 6 | 5 | 11
    Emergency Department | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Skin and Soft Tissue Infection (SSTI)
Description: Recurrence of skin and soft tissue infections at follow up periods (6 weeks, 6 months, and 12 months). At least 1 follow up must be completed.
Time Frame: 12 months
Population: Participants with at least 1 study evaluation at 6 weeks, 6 months, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Number analyzed (Participants) | 5 | 4
Participants | 1 | 2

2. Secondary Outcome: Number of Participants Undergoing Repeat Surgery or Incision/Drainage Procedure for Skin and Soft Tissue Infection
Description: Interval repeat surgery or Incision/Drainage procedure for skin and soft tissue infection assessed at follow up periods (6 weeks, 6 months, and 12 months). At least 1 follow up must be completed.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Number analyzed (Participants) | 5 | 4
Participants | 0 | 2

3. Other Pre Specified Outcome: Participants Who Missed School Due to MRSA SSTI
Description: Parents of participants will be asked whether their child have missed any school days due to MRSA SSTI. Parents will be asked about number of school days missed.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

4. Other Pre Specified Outcome: Mean Adherence to Intervention
Description: Adherence will be reported on a 5 point scale for child and other family members:
  1. - "I always did the hygiene recommendations/bleach baths/mupirocin as recommended".
  2. - "I sometimes didn't do the hygiene recommendations/bleach baths/mupirocin knowingly or unknowingly, but never omitted more than one time/dose/bath in a row"
  3. - "I sometimes didn't do the hygiene recommendations/bleach baths/mupirocin knowingly or unknowingly, but never omitted more than one day/week in a row"
  4. - "I missed hygiene recommendations/bleach baths/mupirocin, knowingly or unknowingly, for two or more days/weeks in a row".
  5. - "I missed most hygiene recommendations/bleach baths/mupirocin, knowingly or unknowingly."
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Number analyzed (Participants) | 5 | 4
score on a scale | 1 (0) | 1.5 (1)

5. Other Pre Specified Outcome: Number of Parents Who Missed Work
Description: frequency of work absences due to child's MRSA infection
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
Number analyzed (Participants) | 5 | 4
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hygiene Education | Hygiene Education and Decolonization
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hygiene Education (N=5) | Hygiene Education and Decolonization (N=4)
Nosebleed (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
We enrolled 14 subjects with only 9 completing at least one outcome assessment. This was far below the 118 (total) or 59/arm needed for appropriate statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02127658/Prot_SAP_000.pdf